CLINICAL TRIAL: NCT07024199
Title: Comparison of the Effectiveness of Paracetamol With Ibuprofen or Paracetamol With Metamizole in Treating Pain in Acute Pancreatitis in Children: a Randomized Trial
Brief Title: Comparison of the Effectiveness of Paracetamol With Ibuprofen or Paracetamol With Metamizole in Treating Pain in Acute Pancreatitis in Children
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, Aleksandra Banaszkiewicz, Prof. Aleksandra Banaszkiewicz, MD, PhD, Medical University of Warsaw
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: APPain
Record Dates: First submitted 2025-02-28; First posted 2025-06-17 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Pancreatitis, Acute; Pain, Acute; Pancreatic Disease; Pancreatic Diseases; Gastroenterology; Pancreatitis; Paediatrics
Keywords: acute pancreatitis; acute pain; painkillers; pancreatitis
MeSH Terms: conditions — Pancreatitis; Acute Pain; Pancreatic Diseases | interventions — Acetaminophen; Ibuprofen; Dipyrone

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Paracetamol + Iburprofen (Experimental): Group A will receive a dose of Paracetamol B. Braun/Paracetamol Kabi intravenously 15 mg/kg body weight (maximum 1000 mg/dose) and Ibuprofen B.Braun/Ibuprofen Kabi intravenously 10 mg/kg body weight (maximum 400 mg/dose).
  Interventions: Other: The initial pain assessment; Drug: Drug administration according to protocol (paracetamol + ibuprofen OR paracetamol + metamizol); Other: The effectiveness of the treatment
- Paracetamol + Metamizol (Experimental): Group B will receive a dose of Paracetamol B. Braun/Paracetamol Kabi intravenously 15 mg/kg body weight (maximum 1000 mg/dose) and Metamizol-SF/Metamizole Kabi/Pyralgin intravenously 15 mg/kg body weight (maximum 100 mg/dose).
  Interventions: Other: The initial pain assessment; Drug: Drug administration according to protocol (paracetamol + ibuprofen OR paracetamol + metamizol); Other: The effectiveness of the treatment

INTERVENTIONS:
Other: The initial pain assessment — The initial pain assessment will be carried out according to pain assessment scales in children adapted to the patient's age and cognitive abilities (NRS, FLACC).
Drug: Drug administration according to protocol (paracetamol + ibuprofen OR paracetamol + metamizol) — Group A will receive a dose of Paracetamol B. Braun/Paracetamol Kabi intravenously 15 mg/kg body weight (maximum 1000 mg/dose) and Ibuprofen B.Braun/Ibuprofen Kabi intravenously 10 mg/kg body weight (maximum 400 mg/dose).
  Group B will receive a dose of Paracetamol B. Braun/Paracetamol Kabi intravenously 15 mg/kg body weight (maximum 1000 mg/dose) and Metamizol-SF/Metamizole Kabi/Pyralgin intravenously 15 mg/kg body weight (maximum 100 mg/dose).
Other: The effectiveness of the treatment — The effectiveness of the treatment will be assessed 60 minutes after the start of the intervention according to pain assessment scales in children adapted to the patient's age and cognitive abilities (NRS, FLACC).

SUMMARY:
The aim of the study is to assess the effectiveness and tolerance of pain treatment in AP in children using intravenous paracetamol in combination with ibuprofen or paracetamol in combination with metamizole. The study is prospective, interventional, and randomized.

DETAILED DESCRIPTION:
Patients with AP diagnosed based on the INSPIRE criteria who meet the inclusion as mentioned above criteria for the study will be randomized (based on a computer-generated randomization list, in blocks of four people) to treatment with one of two regimens:

Group A will receive a dose of paracetamol intravenously 15 mg/kg body weight (maximum 1000 mg/dose) and ibuprofen 10 mg/kg body weight (maximum 400 mg/dose).

Group B will receive a dose of paracetamol intravenously 15 mg/kg body weight (maximum 1000 mg/dose) and metamizole 15 mg/kg body weight (maximum 100 mg/dose).

The initial pain assessment will be carried out according to pain assessment scales in children adapted to the patient's age and cognitive abilities (NRS, Wong-Baker Faces Scale/FLACC- attached). The effectiveness of the treatment will be assessed 60 minutes after the start of the intervention.

Before starting the intervention, all patients during obtaining peripheral intravenous access will undergo a panel of laboratory tests including: alanine aminotransferase, aspartate aminotransferase and gamma-glutamyltransferase activity, total, conjugated and unconjugated bilirubin level, peripheral blood morphology, C-reactive protein, glucose, creatinine, calcium, albumin and urea nitrogen level. Oral and/or intravenous fluid supply in the range of 1.5 to 2 times the daily requirement will be provided, as well as early low-fat enteral nutrition.

After the intervention is completed, the decision on further analgesic treatment will remain at the discretion of the attending physician.

In addition, during the examination, data about the patient will be collected, such as: age, gender, body weight, height, history of chronic diseases and congenital defects, medications taken, reported allergies and family history, with particular emphasis on pancreatic diseases, as well as the results of laboratory tests and imaging, as well as data on possible side effects of the treatment. The patient will be observed for 48 hours from the start of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of AP according to the INSPPIRE mentioned above criteria,
* age from 3 to 18 years of age,
* abdominal pain on admission assessed on the Numerical Rating Scale (NRS) or FLACC >= 4 points,
* no analgesic treatment before enrolment in the study OR the last dose of analgesic drug (paracetamol, ibuprofen, metamizole) taken ≥ 6 hours before enrolment for examination,
* consent of legal guardians and the child (in the case of patients ≥16 years of age) to participate in the study.

Exclusion Criteria - patients:

* who took the last dose of painkiller (paracetamol, ibuprofen, metamizole) < 6 hours before entering the study,
* allergic to acetylsalicylic acid, other NSAIDs, paracetamol, metamizole,
* with inflammatory bowel disease,
* with gastrointestinal bleeding and other active bleeding,
* with gastric and/or duodenal ulcer disease,
* chronically taking paracetamol, NSAIDs, metamizole,
* with liver failure,
* with heart failure according to the NYHA II-IV scale,
* with acute and chronic renal failure,
* with cancer,
* whose legal guardians did not consent to participate in the study,
* who did not consent to participate in the study (applies to patients > 16 years of age).

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in pain intensity assessed at the 60th minute of the examination using ONE of the SCALES. | at the 60th minute after introduction of the intervention
  The number of patients who observed a reduction in pain intensity of <4 points on the NRS scale (for children from 7 years of age) or FLACC scale (for children from 3 to 7 years of age) in both study groups, assessed at the 60th minute of the study.
  NRS is used to assess pain severity at a given moment using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable."
  The FLACC scale [Face, Legs, Activity, Cry, Consolability] is used to assess pain between the ages of 2 months and 7 years or in individuals who are unable to communicate their pain. The scale is scored in a range of 0-10, with 0 representing no pain. The scale has 5 criteria, which are each assigned a score of 0, 1 or 2.

SECONDARY OUTCOMES:
Length of hospitalization. | at the time of discharge (up to 14 days)
  Length of hospitalization in both study groups.
Consumption of opioid drugs. | at the 48th hour after introduction of the intervention
  Consumption of opioid drugs within 48 hours from the start of the study calculated per morphine equivalent/kg body weight.
Reduction in pain intensity assessed at the 6th, 24th and 48th hour. | at 6th, 24th and 48th hour after introduction of the intervention
  The number of patients who observed a reduction in pain intensity by at least 2 points on the NRS scale (for children aged 7 years and over) or FLACC scale (for children aged 3 to 7 years) in both study groups, assessed at 6, 24, and 48 hours of the study.
  NRS is used to assess pain severity at a given moment using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable."
  The FLACC scale [Face, Legs, Activity, Cry, Consolability] is used to assess pain between the ages of 2 months and 7 years or in individuals who are unable to communicate their pain. The scale is scored in a range of 0-10, with 0 representing no pain. The scale has 5 criteria, which are each assigned a score of 0, 1 or 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Paediatric Gastroenterology and Nutrition, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided